CLINICAL TRIAL: NCT00647231
Title: Protocol HKT-500-US12: A Randomized, Multicenter, Double-Blind, Single Dose Study of the Analgesic Properties of HKT-500 and Placebo in Subjects With Pain Caused by Mild to Moderate Osteoarthritis of the Knee
Brief Title: HKT-500-US12 In Adult Patients With OA Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hisamitsu Pharmaceutical Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple
Other Study IDs: HKT-500-US12
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis,Knee,Ketoprofen,Pain,Patch,Analgesic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A, 2, II, HKT-500 Topical Patch (Experimental): A Randomized, Multicenter, Double-Blind, Single Dose Study of the Analgesic Properties of HKT-500 and Placebo in Subjects With Pain Caused by Mild to Moderate Osteoarthritis of the Knee
  Interventions: Drug: HKT-500 Topical Patch
- Placebo Patch (Placebo Comparator): Treatment with placebo patch
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: HKT-500 Topical Patch — Treatment with Ketoprofen Topical Patch
  Other Names: HKT-500; Ketoprofen
  Arms: A, 2, II, HKT-500 Topical Patch
Other: Placebo Patch — Treatment with placebo patch
  Other Names: Sham tratment
  Arms: Placebo Patch

SUMMARY:
The objective of this study is to characterize the analgesic properties of single dose study of HKT-500 in subjects with pain caused by mild to moderate OA of the knee

DETAILED DESCRIPTION:
A Randomized, Multicenter, Double-Blind, Single Dose Study of the Analgesic Properties of HKT-500 and Placebo in Subjects with Pain Caused by Mild to Moderate Osteoarthritis of the Knee

ELIGIBILITY:
Inclusion Criteria:

* male or female 45 years of age or older
* with osteoarthritis of the knee

Exclusion Criteria:

* subject is a woman of childbearing potential
* who has a positive urine pregnancy test,
* is lactating, or who is not surgically sterile

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Time to Onset and Duration | 36 hours

SECONDARY OUTCOMES:
Outcome Time Frame | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Furuta, Study Director — Hisamitsu
Locations (28):
- United States (28):
  - Hisamitsu Investigator Site, Birmingham, Alabama
  - Hisamitsu Investigator Site, Phoenix, Arizona
  - Hisamitsu Investigator Site, Little Rock, Arkansas
  - Hisamitsu Investigator Site, Burbank, California
  - Hisamitsu Investigator Site, Escondido, California
  - Hisamitsu Investigator Site, Northridge, California
  - Hisamitsu Investigator Site, Colorado Springs, Colorado
  - Hisamitsu Investigator Site, DeLand, Florida
  - Hisamitsu Investigator Site, Hallandale, Florida
  - Hisamitsu Investigator Site, Ocala, Florida
  - Hisamitsu Investigator Site, Ormond Beach, Florida
  - Hisamitsu Investigator Site, Austell, Georgia
  - Hisamitsu Investigator Site, Savannah, Georgia
  - Hisamitsu Investigator Site, Stockbridge, Georgia
  - Hisamitsu Investigator Site, Chicago, Illinois
  - Hisamitsu Investigator Site, Madisonville, Kentucky
  - Hisamitsu Investigator Site, Baton Rouge, Louisiana
  - Hisamitsu Investigator Site, Lake Charles, Louisiana
  - Hisamitsu Investigator Site, Flint, Michigan
  - Hisamitsu Investigator Site, Omaha, Nebraska
  - Hisamitsu Investigator Site, Berlin, New Jersey
  - Hisamitsu Investigator Site, Raleigh, North Carolina
  - Hisamitsu Investigator Site, Cincinnati, Ohio
  - Hisamitsu Investigator Site, Zanesville, Ohio
  - Hisamitsu Investigator Site, Oklahoma City, Oklahoma
  - Hisamitsu Investigator Site, Duncansville, Pennsylvania
  - Hisamitsu Investigator Site, Houston, Texas
  - Hisamitsu Investigator Site, Salt Lake City, Utah